CLINICAL TRIAL: NCT00043004
Title: CLOCC Trial (Chemotherapy + Local Ablation Versus Chemotherapy) Randomized Phase II Study Of Local Treatment Of Liver Metastases By Radiofrequency Combined With Chemotherapy Versus Chemotherapy Alone In Patients With Unresectable Colorectal Liver Metastases
Brief Title: Chemotherapy and Bevacizumab With or Without Radiofrequency Ablation in Treating Unresectable Liver Metastases in Patients With Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Arbeitsgruppe Lebermetastasen und Tumoren (Other); Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-40004; EORTC-40004; ALM-CAO-EORTC-40004; NCRI-EORTC-40004
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: liver metastases; stage IV colon cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin; Radiofrequency Ablation

INTERVENTIONS:
Biological: bevacizumab
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin
Procedure: conventional surgery
Procedure: radiofrequency ablation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread by blocking blood flow. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiofrequency ablation uses high-frequency electric current to kill tumor cells. It is not yet known if chemotherapy is more effective with or without radiofrequency ablation in treating liver metastases.

PURPOSE: This randomized phase II trial is studying combination chemotherapy, bevacizumab, and radiofrequency ablation to see how well they work compared to combination chemotherapy and bevacizumab alone in treating unresectable liver metastases in patients with colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the 30-month overall survival rate of patients with unresectable liver metastases secondary to colorectal adenocarcinoma treated with chemotherapy and bevacizumab with or without radiofrequency interstitial ablation.

Secondary

* Compare overall survival of patients treated with these regimens.
* Compare quality of life of patients treated with these regimens.
* Determine the health economics associated with this study.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to treatment center, prior adjuvant chemotherapy for primary cancer (yes vs no), prior chemotherapy for liver metastases (yes vs no), and route of randomization (before surgery vs during surgery). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Within 4 weeks of randomization, patients undergo radiofrequency interstitial ablation (RFA) with or without additional resection of resectable lesions. Within 8 weeks after RFA, patients receive chemotherapy and bevacizumab.
* Arm II: Within 4 weeks of randomization, patients receive chemotherapy and bevacizumab.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Patients in both arms receive one of the following chemotherapy and bevacizumab regimens to be determined by participating center:

* Regimen A: Patients receive oxaliplatin IV over 2 hours on day 1 of weeks 1, 3, and 5 and leucovorin calcium IV over 2 hours followed by fluorouracil IV continuously over 24 hours on day 1 of weeks 1-6 and bevacizumab IV over 30-90 minutes on days 1 or 2, 15 or 16, and 29 or 30. Treatment repeats every 7 weeks for 4 courses.
* Regimen B: Patients receive oxaliplatin IV and leucovorin calcium IV over 2 hours on day 1 followed by fluorouracil IV continuously over 46 hours and bevacizumab IV over 30-90 minutes on day 1 or 3. Treatment repeats every 15 days for 12 courses.
* Regimen C: Patients receive oxaliplatin IV over 2 hours on day 1 and leucovorin calcium IV over 2 hours followed by fluorouracil IV continuously over 22 hours on days 1 and 2 and bevacizumab IV over 30-90 minutes on day 1 or 3. Treatment repeats every 15 days for 12 courses.

Quality of life is assessed at baseline, within 1 week after completion of RFA (arm I only), within 1 week before start of chemotherapy (arm I only), at weeks 6, 12, 18, and 24 during chemotherapy, every 3 months for 2 years after treatment, and then every 6 months thereafter.

After completion of study treatment, patients are followed every 3 months for 2½ years and then every 6 months thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 152 patients (71 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Unresectable liver metastases secondary to colorectal adenocarcinoma, including:

  * Metastases that cannot be radically resected due to size, location, or number of deposits
  * Metastases invading right and left branches of hepatic artery or portal vein
  * Metastases extended to the 3 main hepatic veins
* No detectable extra-hepatic disease
* Fewer than 10 metastatic deposits on liver
* Total metastatic involvement of liver no more than 50%
* Adequate treatment of all metastatic lesions deemed possible either by radiofrequency interstitial ablation (RFA) alone or by a combination of resection of resectable lesions and RFA of the remaining unresectable lesions

  * Maximum diameter of 4 cm for lesions to be treated with RFA
  * No maximum diameter of lesions to be resected as long as negative resection margins are obtainable
* If synchronous liver metastases, must have undergone prior resection of primary tumor

PATIENT CHARACTERISTICS:

Age

* 18 to 80

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* No bleeding disorder or coagulopathy or need for full-dose anticoagulation

Hepatic

* Bilirubin less than 3 times upper limit of normal (ULN)
* Alkaline phosphatase less than 3 times ULN

Renal

* Creatinine less than 2 times ULN
* Protein < 0.5 g/24 hr urine collection if proteinuria positive by dipstick

Cardiovascular

* No uncontrolled congestive heart failure
* No uncontrolled angina pectoris
* No uncontrolled hypertension
* No uncontrolled arrhythmia
* No myocardial infarction within the past 12 months
* No cerebrovascular accident or transient ischemic attack within the past 6 months

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No greater than grade 1 peripheral neuropathy
* No significant neurologic or psychiatric disorder
* No active infection
* No contraindication to the use of fluorouracil, leucovorin calcium, oxaliplatin, or bevacizumab
* No other malignancy within the past 10 years except nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy except for metastatic disease confined to the liver

  * Prior fluorouracil, leucovorin calcium, and oxaliplatin allowed if administered for at least 3 courses (2 weeks each) but no longer than 3 months with at least stabilization of disease achieved
* Prior adjuvant chemotherapy for primary cancer allowed except for patients who received oxaliplatin and have been diagnosed with metastatic disease within 12 months after completion of adjuvant treatment

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* More than 28 days since major surgery or open biopsy past 28 days
* More than 28 days since significant traumatic injury

Other

* No other concurrent investigational treatment
* No other concurrent anticancer therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2002-05; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Survival rate as measured by Kaplan Meier method at 30 months

SECONDARY OUTCOMES:
Overall survival as measured by Logrank every 3 months for 30 months then every 6 months thereafter
Progression-free survival as measured by Logrank every 3 months for 30 months then every 6 months thereafter
Toxicity as measured by CTC version 2.0 every 3 months for 30 months then every 6 months thereafter
Quality of life as measured by Quality of Life Questionnaire Core 30 (QLQ-C30) version 3.0 at baseline, weeks 6, 12, 18, and 24, every 3 months for years 1-2 after start of treatment, then every 6 months thereafter
Response to treatment (arm II) as measured by RECIST criteria from start of treatment until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Theo Ruers, MD, Study Chair — Universitair Medisch Centrum St. Radboud - Nijmegen; Wolf O. Bechstein, MD, Study Chair — Arbeitsgruppe Lebermetastasen und Tumoren; Jonathan A. Ledermann, MD, Study Chair — Cancer Research UK
Locations (43):
- Allgemeines Krankenhaus - Universitatskliniken, Vienna, Austria
- Belgium (5):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Clinique Universitaire De Mont-Godinne, Mont-Godinne Yvoir
- National Cancer Institute - Cairo, Cairo, Egypt
- France (4):
  - Centre Hospitalier Regional et Universitaire d'Angers, Angers
  - Centre Hospitalier Universitaire Ambroise Pare - Boulogne, Boulogne-Billancourt
  - Hopital Universitaire Hautepierre, Strasbourg
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
- Germany (5):
  - Robert Roessle Comprehensive Cancer Center at University of Berlin - Charite Campus Buch, Berlin
  - Kliniken Essen - Mitte, Essen
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Staedtische Kliniken Frankfurt am Main - Hoechst, Frankfurt
  - Klinikum der Universitaet Regensburg, Regensburg
- National Institute of Oncology, Budapest, Hungary
- Azienda Ospedaliera S. Camillo-Forlanini, Rome, Italy
- Netherlands (10):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Amphia Ziekenhuis - locatie Langendijk, Breda
  - Medisch Spectrum Twente, Enschede
  - Atrium Medical Centre - Heerlen, Heerlen
  - Medisch Centrum Leeuwarden - Zuid, Leeuwarden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - University Medical Center Utrecht, Utrecht
  - Maxima Medisch Centrum - Veldhoven, Veldhoven
- Sweden (3):
  - Sahlgrenska University Hospital at Gothenburg University, Gothenburg (Goteborg)
  - Karolinska University Hospital - Huddinge, Stockholm
  - Uppsala University Hospital, Uppsala
- United Kingdom (12):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Leicester General Hospital, Leicester, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Cancer Research UK and University College London Cancer Trials Centre, London, England
  - University College of London Hospitals, London, England
  - Manchester Royal Infirmary, Manchester, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Churchill Hospital, Oxford, England
  - Royal South Hants Hospital, Southampton, England
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Glan Clywd District General Hospital, Rhyl, Denbighshire, Wales

REFERENCES:
- [Result] Ruers T, van Coevorden F, Pierie J, et al.: Radiofrequency ablation (RFA) combined with chemotherapy for unresectable colorectal liver metastases (CRC LM): interim results of a randomised phase II study of the EORTC-NCRI CCSG-ALM Intergroup 40004 (CLOCC). [Abstract] J Clin Oncol 26 (Suppl 15): A-9535, 2008.
- [Derived] Ruers T, Punt C, Van Coevorden F, Pierie JPEN, Borel-Rinkes I, Ledermann JA, Poston G, Bechstein W, Lentz MA, Mauer M, Van Cutsem E, Lutz MP, Nordlinger B; EORTC Gastro-Intestinal Tract Cancer Group; Arbeitsgruppe Lebermetastasen und-tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie (ALM-CAO) and the National Cancer Research Institute Colorectal Clinical Study Group (NCRI CCSG). Radiofrequency ablation combined with systemic treatment versus systemic treatment alone in patients with non-resectable colorectal liver metastases: a randomized EORTC Intergroup phase II study (EORTC 40004). Ann Oncol. 2012 Oct;23(10):2619-2626. doi: 10.1093/annonc/mds053. Epub 2012 Mar 19. PMID 22431703